CLINICAL TRIAL: NCT06640764
Title: Étude Prospective, Multicentrique, Non contrôlée, Non randomisée, Ouverte évaluant la Performance et la stabilité de l'Implant fémoral Non cimenté SMS
Brief Title: Multicentre SMS Study - FR
Status: Recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P01.019.07
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Dysplasia of Hip Joint; Hip Osteoarthritis; Traumatic Arthritis of Hip; Avascular Necrosis of Femur Head
MeSH Terms: conditions — Osteoarthritis, Hip; Femur Head Necrosis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Total Hip Arthroplasty — Total Hip Arthroplasty with SMS Femoral Stem (Medacta)

SUMMARY:
Prospective, multicentre, non controled, non randomised, clinical study to assess the performance and the stability of SMS femoral stem

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from a severely painful and/or disabling hip joint due to osteoarthritis, traumatic arthritis, developmental dysplasia of the hip, or avascular necrosis of the femoral head, and requiring a total hip replacement.
* Patient who will receive a Medacta SMS femoral stem.
* Patient agrees to comply with the study requirements.
* Patient has signed the consent form.
* Patient is affiliated with a social security system.
* Patient aged 18 to 75 years

Exclusion Criteria:

* Participation in biomedical research.
* Minor patient.
* Protected adult patient.
* Vulnerable individuals as defined by Article L1121-6 of the Public Health Code.
* Pregnant or breastfeeding women.
* Patient unable to express their non-opposition.
* Patient refusing the collection of their personal data.
* Acute, systemic, or chronic infection. Skeletal immaturity.
* Grossly deformed anatomy (at the surgeon's discretion).
* Osteomalacia for which the fixation of an uncemented implant is contraindicated.
* Patient suffering from active rheumatoid arthritis or osteoporosis.
* Patient with metabolic disorders likely to impair bone formation when the fixation of an uncemented implant is contraindicated.
* Patient suffering from muscle atrophy or neuromuscular disease.
* Patient with an allergy to the implant material.
* Any patient who cannot or does not wish to give their informed consent to participate in the study.
* Patient whose prospects of regaining independent mobility would be compromised by known coexisting medical problems.
* Any contraindication mentioned in the instructions for use of the investigational medical device.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from a severely painful and/or disabling hip joint (osteoarthritis, traumatic arthritis, developmental dysplasia of the hip, avascular necrosis of the femoral head) requiring a total hip prosthesis and who will receive a Medacta SMS femoral stem.
  Patients will be able to participate in other non-interventional research for the duration of the study.
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2034-09-01 (Estimated); Study Completion 2037-09-01 (Estimated)

PRIMARY OUTCOMES:
Survival rate of SMS femoral stem | From enrollment to the end of treatment at 10 years
  Survival analysis accordin to the Kaplan-Meier method

SECONDARY OUTCOMES:
Evaluation of the clinical performance of the SMS femoral stem | From enrollment to the end of treatment at 10 years
  Clinical performance of the SMS femoral stem evaluated through the Harris Hip Score. The Harris Hip Score is a standardized measure used to assess the severity of hip pain and functional limitations in individuals with hip conditions. The maximum score possible is 100. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.
Evaluation of the hip function | From enrollment to the end of treatment at 10 years
  Hip function evaluated through the Oxford Hip Score. The Oxford Hip Score (OHS) is a short 12-item patient-reported PRO specifically designed and developed to assess function and pain with patients undergoing hip replacement surgery. The total gives a minimum score of 12 and a maximum of 60. A higher score implies a greater degree of disability.
Evaluation of the quality of life | From enrollment to the end of treatment at 10 years
  Quality of life evaluated through the EuroQol Score (EQ-5D-5L). The EQ-5D family of instruments has been developed to describe and value health across a wide range of disease areas. Each EQ-5D instrument comprises a short descriptive system questionnaire and a visual analogue scale (EQ VAS) that are cognitively undemanding, taking only a few minutes to complete. The questionnaire provides a simple descriptive profile of a respondent's health state. The EQ VAS provides an alternative way to elicit an individual's rating of their own overall current health
Evaluation of the safety (adverse events) of the SMS femoral stem | From enrollment to the end of treatment at 10 years
  Safety of the SMS femoral stem evaluated through the collection of the intraoperative and postoperative complications
Evaluation of the stability and the fixation of the SMS femoral stem | From enrollment to the end of treatment at 10 years
  Stability and fixation of the SMS femoral stem evaluated through the radiographic anaysis, assessing the position of the implant (subsidence and migration), the presence of radiolucent lines, the implant breakage.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de l'Union, Saint-Jean, France